CLINICAL TRIAL: NCT01294657
Title: Obesity: Cancer Risk Among African Americans-Developing Interventions Through Community Collaboration
Brief Title: Obesity: Cancer Risk Among African Americans
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Other Study IDs: 2010-0161
Record Dates: First submitted 2011-02-10; First posted 2011-02-11 (Estimated); Last update posted 2019-05-10 (Actual); Status verified 2019-05

CONDITIONS: Cancer; Obesity
Keywords: Obesity; Cancer Risk; African Americans; Diet; Physical Activity
MeSH Terms: conditions — Neoplasms; Obesity; Motor Activity | interventions — Surveys and Questionnaires; Counseling

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 16 saliva samples to be collected for hormone testing.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- HE Group: Health Education [HE] - Counseling, referrals to resources + self-help materials; 2 HE interventions at Baseline + 6 month visits.
  Interventions: Behavioral: Health Education
- MAPS Group: Motivation And Problem Solving (MAPS) - HE + 12 telephone counseling sessions over 1-year period (average 1 call/month).
  Interventions: Behavioral: Health Education; Behavioral: MAPS

INTERVENTIONS:
Behavioral: Health Education — Counseling, referrals to available resources and self-help materials on Day 1, at 6 and 12 month visits, along with surveys at 6 and 12 months.
  Other Names: Survey; Counseling
Behavioral: MAPS — 12 counseling phone calls over 1 year, lasting about 20-30 minutes.
  Other Names: Counseling
  Groups: MAPS Group

SUMMARY:
The goal of this research study is to learn if a motivation and problem solving (MAPS) program can help improve diet and levels of physical activity in African Americans who are overweight.

DETAILED DESCRIPTION:
Day 1 Study Visit:

If you are found eligible to take part in this study, the following tests and procedures will be performed on Day 1 (the same day you complete the screening tests and sign this consent form):

* You will complete a computer-based survey about your mood, diet, and physical activity. The survey should take about 90 minutes total to complete.
* Your blood pressure will be measured.
* Your height, weight, and waistline will be measured. To measure your waistline accurately, you may be asked to lift your shirt to expose your stomach area and to lower your pants to expose your mid-hip area. Waistline measurements will only take about 10 minutes to complete and will be performed in a private area.
* Your non-fasting blood glucose and cholesterol levels will be measured (with 2 small finger pricks).
* You will be asked to provide a 7-day record of your physical activity using a small device called an accelerometer. The accelerometer will be worn on your hip and measures the amount of physical activity you do. You will be given a prepaid envelope to return the accelerometer to the study staff.

Study Groups and Study Procedures:

At the Day 1 study visit, you will be randomly assigned (as in the flip of a coin) into 1 of 2 study groups.

If you are in Group 1 or 2, you will receive health education on Day 1, 6 months, and 12 months later. Health education includes:

* A brief counseling session with a study staff member to talk about diet and your physical activity levels
* Referrals to available resources for help with your diet and physical activity
* Self-help materials that are designed to help you learn how to improve your diet and physical activity

At Months 6 and 12, you will also:

* Complete the computer-based survey about your mood, diet, and physical activity.
* Have your height, weight, waistline and blood pressure measured.
* Your non-fasting blood glucose and cholesterol levels will be measured.
* Be given an accelerometer to wear for 7 days.You will be given a prepaid envelope to return the accelerometer to the study staff.

If you are in Group 2, you will also take part in the MAPS program. For the MAPS program, you will have 12 counseling phone calls over 1 year. Each of these phone calls will be digitally recorded and should last about 20-30 minutes. You may decline to have your counseling phone call recorded if it makes you feel uncomfortable. The purpose of the phone calls are to provide support to you on changes in your diet or physical activity and to answer any questions you may have about your program.

Length of Study:

You will remain on the study for up to 1 year. Your participation on this study will be over once you complete the study visit at Month 12.

Other Important Information:

You may be contacted by phone, mail, and/or email at any time while you are taking part in this study to be reminded about the study visits. You will be asked to give the names and contact information for family members and/or friends for the study staff to contact in the event there is trouble reaching you first.

If the accelerometer is lost or stolen, you will not be responsible for the replacement cost, but you should tell the study staff right away.

All participant's paper files will be stored in locked file cabinets and all data files will be stored in a password-protected databases. The information discussed during the counseling phone calls will be kept confidential. Only members of the research team will have access to the recordings.

This is an investigational study.

Up to 300 participants will take part in this study. All will be enrolled at MD Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Self-reported African American race
2. Ability to engage in low to moderate physical activity as determined by the Physical Activity Readiness Questionnaire (PAR-Q) or by physicians clearance (letter from physician or nurse practitioner) if currently taking medication for blood pressure or diabetes.
3. Blood pressure reading <140/90 mm Hg or by physicians clearance (letter from physician or nurse practitioner) if blood pressure reading >=140/90 mm Hg.
4. Functioning telephone number
5. 18-65 years of age
6. Overweight or obese as defined by BMI
7. Not currently exercising (<150 minutes/week) and/or not consuming 5 or more servings of fruits and vegetables per day

Exclusion Criteria:

1. Pressure readings >140/90 mm Hg, as defined by the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure, will be excluded from the study.
2. Currently taking medication for blood pressure or heart condition, or other physical limitations that might be aggravated by participation in moderate-intensity PA as measured using the PA Readiness Questionnaire, and any physical limitation that prevents engaging in PA.
3. Pregnant or thinking about becoming pregnant during the study period
4. Another household member enrolled in the study
5. Member of the church advisory board

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: African Americans will be recruited from Windsor Village United Methodist Church in Houston, Texas.
Sampling Method: Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2011-01 (Actual); Primary Completion 2020-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Efficacy of a Motivation and Problem Solving (MAPS) Approach to Promoting and Facilitating Positive Health Behavior Change Among African Americans | 6 months
  Effects of MAPS on each of modifiable risk factors, assessed at 6 and 12-month follow-up visits using, using Questionnaire Design System (QDS), a computer-administered self-interview format.

CONTACTS AND LOCATIONS:
Overall Officials: Lorna H. McNeill, PHD,MPH, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org